CLINICAL TRIAL: NCT07384741
Title: L'Utilizzo Della realtà Virtuale Mediante l'Impiego Del Visore Ottico Nel Paziente Oncologico Sottoposto al Posizionamento di PICC e PICC-PORT
Brief Title: Using Virtual Reality During PICC and PICC-PORT Placement in Cancer Patients
Acronym: VR-PICCPORT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Principal Investigator, Paola Tiatto, Coordinatrice Infermieristica U.O. Anestesia e Rianimazione IOV Sede di Castelfranco Veneto, Istituto Oncologico Veneto IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-18; Ministero della Salute (Other: Ministero della Salute - ricerca corrente)
Record Dates: First submitted 2026-01-16; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Neoplams; Anxiety; Pain; Satisfaction; Peripherally Inserted Central Catheters; Catheterization, Central Venous
Keywords: virtual reality; cancer patient; PICC; PICC-PORT; anxiety; pain; satisfaction
MeSH Terms: conditions — Anxiety Disorders; Pain; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Virtual reality + Standard of care (VR+SOC) (Experimental): Patients will receive standard care for PICC or PICC-PORT placement, combined with VR delivered via a head-mounted display throughout the procedure.The VR system used is HypnoVR, developed by Medival s.r.l. and include a VR headset, Lenovo tablet, and Bluetooth headphones.
  HypnoVR integrates clinical hypnosis with immersive virtual environments, guided breathing, music therapy-based compositions, and cardiac coherence techniques, providing multisensory therapeutic immersion. Continuous communication with patients will be maintained throughout the session, and patients may select preferred visual and musical environments.
  Interventions: Device: Virtual reality VR
- Arm B: Standard of Care (SOC) (No Intervention): Patients will undergo standard care for PICC or PICC-PORT placement without VR.

INTERVENTIONS:
Device: Virtual reality VR — Patients will receive standard care for PICC or PICC-PORT placement, combined with VR (Hypno VR) delivered via a head-mounted display throughout the procedure. HypnoVR integrates clinical hypnosis with immersive virtual environments, guided breathing, music therapy-based compositions, and cardiac coherence techniques, providing multisensory therapeutic immersion. Continuous communication with patients will be maintained throughout the session, and patients may select preferred visual and musical environments.
  Arms: Arm A: Virtual reality + Standard of care (VR+SOC)

SUMMARY:
Virtual reality (VR) has increasingly been explored in medical settings as a non-pharmacological intervention for the management of pain and anxiety associated with invasive procedures. By providing immersive and interactive environments, VR is thought to modulate both sensory and emotional components of pain through mechanisms involving focused attention, cognitive engagement, and altered perception, which share similarities with hypnosis-based approaches. Evidence from previous studies, initially conducted mainly in paediatric populations and more recently extended to adults, suggests that VR may effectively reduce procedural anxiety and pain without increasing procedural duration or clinical workload.

Oncology patients undergoing the placement of vascular access devices, such as peripherally inserted central catheters (PICC) and PICC-PORTs, frequently experience procedural distress, including anxiety and discomfort, related to the invasive nature of the intervention. Procedural anxiety may negatively influence patient experience, cooperation, and overall tolerance of the procedure, potentially increasing the need for pharmacological anxiolytic or analgesic support. Identifying effective, safe, and easily applicable non-pharmacological strategies to reduce distress during these procedures represents a relevant clinical goal in oncology care.

The present study aims to evaluate the effectiveness of virtual reality delivered via a head-mounted display in reducing patient-reported anxiety and pain in adult oncology patients undergoing PICC or PICC-PORT insertion.

This study is designed as a prospective, interventional, randomised controlled trial with a 1:1 allocation ratio using a random number generator within REDCap. A total of 120 patients will be enrolled at a single centre, the Istituto Oncologico Veneto (IRCCS), and randomly assigned to one of two study arms. Participants allocated to the intervention arm will receive VR in addition to the standard of care (VR + SOC) throughout the vascular access placement procedure, while participants in the control arm will undergo the standard procedure alone (SOC).

The VR intervention will be delivered using HypnoVR, a software-based medical device classified as Class I, non-sterile, and compliant with Regulation (EU) 2017/745 on Medical Devices. The intervention will be administered via a head-mounted display with audiovisual content designed to promote relaxation, focused attention, and emotional regulation during the procedure.

The primary outcome measure is the reduction of anxiety levels at the end of the procedure, assessed using the validated Visual Analogue Scale for Anxiety (VAS-A). Secondary outcomes include patient-reported pain, qualitative assessment of procedural comfort, and perceived ease of procedural management as reported by healthcare staff.

Data collection will include both quantitative and qualitative measures within a mixed-methods framework. Quantitative data will be analysed using descriptive and inferential statistical methods to assess differences between study groups, while qualitative data derived from semi-structured interviews will be analysed using the Van Kaam phenomenological method to explore patients' lived experiences. The study aims to provide evidence on the role of virtual reality as a supportive, non-pharmacological option for anxiety and pain management during vascular access placement in oncology patients.

DETAILED DESCRIPTION:
BACKGROUND

In recent years, virtual reality (VR) has found increasingly widespread and innovative applications in the field of medicine, particularly within rehabilitation pathways, medical education, and the management of mental health conditions as well as chronic and acute pain. Numerous studies have demonstrated that the immersive experience created by VR restricts individuals' cognitive capacity to process acute pain and anxiety, and that this approach is more effective than simpler distraction-based methods.

The modulation of anxiety and pain through the use of VR is enabled by mechanisms associated with hypnosis, attentional shifting, and skills acquisition. Hypnosis aims to divert patients' attention away from painful and anxiety-provoking stimuli by immersing them in a virtual environment. The sensory and cognitive hypnotic mechanisms offered by VR lead to diversion of pain signals and interference with their processing at the level of the neuromatrix. Distraction represents a dispersion of attention towards multiple, uncontrolled stimuli, reducing voluntary attentional capacity; in contrast, hypnosis is characterised by a state of focused attention and heightened suggestibility, in which individuals remain conscious while intentionally directing their internal focus. Relaxing virtual environments are capable of modulating emotional responses, reducing both pain and anxiety, while active engagement enhances perceived control and further decreases pain perception. VR is able to influence brain activity by modulating neuromatrix responses to pain and by providing an integrated experience capable of acting across multiple dimensions.

Anxiety and pain are among the most frequently reported sensations before and during vascular access placement, in both paediatric and adult populations. However, the majority of existing literature focuses on the use of VR as a non-pharmacological distraction technique primarily in paediatric patients, largely neglecting its application in adult patients undergoing similar procedures.

The use of VR delivered through a head-mounted display during vascular access placement, specifically PICC and PICC-PORT insertion, in adult populations is only marginally reported in the literature. A prospective, multicentre, randomised controlled study demonstrated reductions in anxiety and pain among patients exposed to VR compared with standard care, without prolonging procedural time and with a reduction in the use of anaesthetic and analgesic agents. However, this study also highlighted that several factors influence patients' responses and the applicability of VR. Individual characteristics such as mood, personality, expectations, and previous experiences may affect responsiveness to VR. Nevertheless, VR represents a valid and promising non-pharmacological alternative for procedural sedation.

RESEARCH QUESTION Is the use of virtual reality delivered through a head-mounted display, worn by oncology patients during vascular access placement, specifically PICC and PICC-PORT, effective in improving the lived procedural experience in terms of anxiety and pain, compared with patients undergoing the standard device implantation procedure? PRIMARY OBJECTIVE The primary objective of the study is to evaluate the effectiveness of virtual reality delivered through a head-mounted display in oncology patients undergoing vascular access placement, specifically PICC and PICC-PORT insertion.

SECONDARY OBJECTIVES

The secondary objectives are as follows:

To evaluate the effectiveness of VR delivered through a head-mounted display in achieving a statistically significant reduction in patient-reported anxiety levels at the end of the procedure compared with the control group.

To evaluate the effectiveness of VR in reducing patient-reported pain levels. ENDPOINTS The primary efficacy endpoint is the success rate of VR, defined as the percentage of patients undergoing PICC or PICC-PORT placement with VR who show a statistically significant reduction in anxiety levels at the end of the procedure compared with patients receiving standard care. Additional outcomes include a more favourable qualitative evaluation of procedural comfort, a potential reduction in perceived pain, and easier procedural management by healthcare staff following PICC or PICC-PORT insertion, compared with the control arm.

STUDY DESIGN Prospective, interventional, randomised controlled study. Randomisation will be performed using REDCap software through a computer-generated random number sequence with a 1:1 allocation ratio.

SAMPLE

A total of 120 patients will be enrolled and allocated to two treatment arms:

Arm A (60 patients): VR delivered via head-mounted display plus standard of care in oncology patients undergoing PICC or PICC-PORT insertion.

Arm B (60 patients): Standard care alone for oncology patients undergoing PICC or PICC-PORT placement.

INCLUSION CRITERIA Age ≥ 18 years Ability to understand the Italian language Oncological diagnosis Patients undergoing PICC or PICC-PORT insertion EXCLUSION CRITERIA Refusal to participate Inability to provide informed consent Visual or auditory impairments Sensory deficits affecting the procedural area Cognitive or psychiatric disorders that could compromise data reliability STUDY DURATION Start of recruitment: 01/07/2025 End of recruitment: 30/04/2026 Data analysis period: 01/05/2026 - 31/07/2026 End of study: 31/07/2026 Total study duration: 12 months STUDY CENTRE The study will be conducted at a single centre: Istituto Oncologico Veneto, within the facilities dedicated to vascular access placement in the Department of Oncological Surgery.

INTERVENTION Arm A: Virtual Reality + Standard of Care (VR + SOC) Patients will receive standard care for PICC or PICC-PORT placement, combined with VR delivered via a head-mounted display throughout the procedure.

The VR system used is HypnoVR, developed by Medival s.r.l. It is a Class I non-sterile software-based medical device compliant with Regulation (EU) 2017/745 on Medical Devices. Accessories compliant with Directive 2014/53/EU include a VR headset, Lenovo tablet, and Bluetooth headphones. The full system is contained in a dedicated transport case. HypnoVR has been marketed in Italy since 2023 and does not contain latex or phthalates.

HypnoVR integrates clinical hypnosis with immersive virtual environments, guided breathing, music therapy-based compositions, and cardiac coherence techniques, providing multisensory therapeutic immersion. Continuous communication with patients will be maintained throughout the session, and patients may select preferred visual and musical environments. HypnoVR can be used in individuals aged seven years and above and is applied across multiple clinical settings, including oncology procedures and vascular access placement.

Arm B: Standard of Care (SOC) Patients will undergo standard care for PICC or PICC-PORT placement without VR. SAMPLE SIZE CALCULATION Primary outcomes selected for sample size calculation were anxiety measured using the VAS-A scale (0-10) and pain measured using the VAS (0-10). Based on literature evidence, physiological parameters such as heart rate and blood pressure were excluded due to multiple confounding factors.

Assumptions included a minimal clinically relevant difference of 1.5 points, an expected standard deviation of 2.5 (Cohen's d = 0.6), a significance level of 0.05 (two-tailed), and a statistical power of 90%. Using the standard formula for comparison of independent means, a sample size of 59 patients per group (118 total) was obtained. Accounting for an anticipated dropout rate of 10%, the final target sample size was set at 120 patients.

DATA COLLECTION Data collection will follow a mixed-methods research design, incorporating both quantitative and qualitative variables. Data will be collected at two time points: before device placement (T0) and after placement (T1).

DATA ANALYSIS Quantitative data will be analysed using descriptive statistics, regression models, and tests of independence to assess associations between independent and outcome variables. Qualitative data derived from semi-structured interviews will be analysed using the Van Kaam method.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18 years or older
* Diagnosis of neoplastic disease (solid or haematological malignancy)
* Patients scheduled for peripherally inserted central catheter (PICC) or PICC-PORT placement
* Ability to understand the Italian language
* Ability and willingness to provide written informed consent

Exclusion Criteria

* Refusal to participate in the study
* Inability to provide informed consent
* Visual or auditory impairments that may interfere with the use of a virtual reality head-mounted display
* Sensory deficits involving the anatomical area affected by the procedure
* Cognitive, neurological, or psychiatric disorders that may compromise comprehension, cooperation, or reliability of patient-reported outcomes
* Any condition judged by the investigator to make participation unsafe or inappropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety (VAS-A, 0-10) from pre-procedure to post-procedure | Baseline (pre-procedure, same day) and immediately after PICC/PICC-PORT placement (end of procedure, same day).
  The change in anxiety score (VAS-A) is calculated as the difference between the post-procedure and pre-procedure values. Positive change scores indicate an increase in anxiety, and negative change scores indicate a decrease.
Change in pain (VAS, 0-10) from pre-procedure to post-procedure | Baseline (pre-procedure, same day) and immediately after the procedure (end of procedure, same day).
  The change in pain score (VAS) is calculated as the difference between the post-procedure and pre-procedure values. Positive change scores indicate an increase, and negative change scores indicate a decrease.
Patient comfort (1-4 Likert) | Immediately after the procedure (end of procedure, same day).
  Single-item rating of comfort during procedure (1=not at all to 4=very)

SECONDARY OUTCOMES:
Perceived helpfulness of intervention (1-4 Likert) | Immediately after the procedure (end of procedure, same day).
  Perceived helpfulness of the intervention will be measured using a study-developed 4-point Likert scale (1 = not at all helpful; 4 = very helpful). Higher scores indicate greater perceived helpfulness.
Change in heart rate (beats per minute) from baseline to end of procedure | Baseline (pre-procedure, same day) and end of procedure (same day).
  Descriptive/exploratory outcome due to potential confounding. Higher values indicate higher heart rate. Unit of Measure: beats per minute (bpm)
Change in mean arterial pressure (mmHg) from baseline to end of procedure | Baseline (pre-procedure, same day) and end of procedure (same day).
  Descriptive/exploratory outcome due to potential confounding. Higher values indicate higher arterial pressure. Unit of Measure: millimeters of mercury (mmHg)
Qualitative Interview | From 24 to 48 hours after the procedure.
  Semi-structured thematic interview exploring patient experience, anxiety, and pain related to the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto (IOV) c/o Ospedale San Giacomo, Via dei Carpani, 16/Z, 31033 Castelfranco Veneto (TV)., Castelfranco Veneto, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data collected during this study will not be shared publicly. Only aggregated and anonymised data will be reported in scientific publications and presentations. Any data sharing beyond these outputs would require additional ethical approval and amendments to the informed consent.

REFERENCES:
- [Result] Ericsson I, Thilander B. Orthodontic relapse in dentitions with reduced periodontal support: an experimental study in dogs. Eur J Orthod. 1980;2(1):51-7. No abstract available. PMID 6935058
- [Result] Basak T, Duman S, Demirtas A. Distraction-based relief of pain associated with peripheral intravenous catheterisation in adults: a randomised controlled trial. J Clin Nurs. 2020 Mar;29(5-6):770-777. doi: 10.1111/jocn.15131. Epub 2019 Dec 16. PMID 31793099
- [Result] Schaake R, Leopold I, Sandberg A, Zenk B, Shafer L, Yu D, Lu X, Theingi S, Udongwo A, Cohen GS, Maresky HS. Virtual Reality for the Management of Pain and Anxiety for IR Procedures: A Prospective, Randomized, Pilot Study on Digital Sedation. J Vasc Interv Radiol. 2024 Jun;35(6):825-833. doi: 10.1016/j.jvir.2024.03.004. Epub 2024 Mar 12. PMID 38484911
- [Result] Ahmadpour N, Randall H, Choksi H, Gao A, Vaughan C, Poronnik P. Virtual Reality interventions for acute and chronic pain management. Int J Biochem Cell Biol. 2019 Sep;114:105568. doi: 10.1016/j.biocel.2019.105568. Epub 2019 Jul 12. PMID 31306747